CLINICAL TRIAL: NCT07312708
Title: LEan Body Mass Development in CriTically Ill Patients, Obtained by bioelectRical impEdance Analysis: a Combined Retrospective and Prospective Observational Cohort Study
Brief Title: Protein Dosing Strategies in Critically Ill Patients: Comparing Actual Body Weight and Fat-Free Mass Approaches in an Observational Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Gelderse Vallei Hospital (Other)
Responsible Party: Principal Investigator, ARH van Zanten, MD PhD, Principal Investigator, Gelderse Vallei Hospital
Other Study IDs: 2403-017
Record Dates: First submitted 2025-12-05; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-10

CONDITIONS: Critical Illness
Keywords: proteins; critical illness; lean body mass; fat free mass; BIA
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ABW fed: This group received proteins based on 1.5 grams per kilogram actual body weight
- FFM fed: This group received proteins based on 1.85 grams per kilogram fat free mass (BIA determined)

SUMMARY:
This study investigates how different methods of calculating protein intake affect recovery and muscle preservation in critically ill patients in the Intensive Care Unit (ICU). Protein is essential for maintaining muscle strength, supporting healing, and improving recovery during critical illness.

At Hospital Gelderse Vallei, patients admitted to the ICU received protein based on actual body weight until 2023; more recently, protein prescriptions have been based on fat-free mass. Bioelectrical impedance analysis (BIA) has been part of standard clinical practice in the ICU since April 2020, meaning that all patients admitted since then have been screened for inclusion in the study.

This design allows for comparison between two groups: one group receiving protein based on actual body weight according to current clinical guidelines (1.5 g/kg body weight), and another group whose protein intake is calculated based on lean body mass (LBM) measured by BIA. BIA measurements are repeated during the ICU stay to monitor changes in body composition.

A total of 310 patients admitted to the ICU between the start of BIA implementation in April 2020 and the transition to fat-free mass-based dosing in 2023 were identified. To allow for balanced comparison, an equal number of 310 patients from the subsequent period, in which protein dosing was based on fat-free mass, were included in the study.

The study compares these two groups to determine whether calculating protein requirements based on lean body mass leads to better clinical outcomes-such as improved recovery (lower mortality and shorter hospital stay), preservation of muscle mass, and lower UCR-than the traditional method based on actual body weight. The data analysis plan was established prior to completion of patient inclusion and database lock.

DETAILED DESCRIPTION:
Patients were enrolled through an opt-out procedure using an information leaflet included in the admission folder. The acquisition of informed consent from patients admitted between April 2020 and July 2023 was deemed neither necessary nor feasible, as the study relies on an anonymized database and no additional measurements are performed. Therefore, the internal committee for research evaluation approved the waiver of informed consent for these patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* a BIA measurement available within 48 hours after ICU admission
* at least one follow-up BIA measurement during ICU stay.

Exclusion Criteria:

* transfer from another ICU resulting in the first BIA measurement >48 hours after admission to GVH
* a previous ICU admission within 2 weeks before the current admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients
Sampling Method: Probability Sample
Enrollment: 620 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | Mortality, defined as death from any cause, from ICU admission until 90 days post-admission
  Short (ICU and 30-day mortality) and long-term mortality (90 days)

SECONDARY OUTCOMES:
ICU and hospital length of stay | From ICU admission until the date of ICU discharge or the documented date of death from any cause, whichever comes first, assessed up to 52 weeks after ICU admission
  Duration of ICU and hospital length of stay in days
Duration of invasive mechanical ventilation (IMV) | Number of days on invasive mechanical ventilation (IMV), defined as the total number of days with IMV from initiation until ICU discharge, assessed up to 52 weeks after ICU admission
  Duration of invasive mechanical ventilation in days
Urea-creatinine ratio during ICU stay | All UCR measurements taken during the ICU stay, from ICU admission to ICU discharge, with each measurement recorded daily and specified by the day relative to ICU admission, up to a maximum of 52 weeks
  Differences in urea-to-creatinine-ratio between both groups during ICU stay
Changes in BIA parameters over time (in kg) | All BIA measurements during the ICU stay, including dry fat-free mass, skeletal muscle mass and fat mass, recorded daily from ICU admission to ICU discharge, up to 52 weeks.
  Changes in BIA (bioelectric impedance analysis) parameters, including fat free mass, sketetal mass and fat mass (all in kg)
Changes in BIA water parameters over time (in L) | All BIA measurements during the ICU stay, such as intracellular water, extracellular water, and total body water, recorded daily from ICU admission to ICU discharge, up to 52 weeks
  Changes in BIA water (bioelectric impedance analysis) parameters in liters
Changes in BIA phase angle | All BIA measurements during the ICU stay, such as phase angle, recorded daily from ICU admission to ICU discharge, up to 52 weeks
  Changes in BIA phase angle

OTHER OUTCOMES:
Protein intake during ICU stay | Daily intake for the first 14 days since ICU admission, or all days on the ICU if this is less than 14 days
  Daily and cumulative (during the first 14 days) protein intake during ICU stay
Energy intake during ICU stay | Daily energy intake for the first 14 days since ICU admission, per day, of all days of ICU stay if ICU stay is shorter than 14 days
  Daily and cumulative (during the first 14 days) energy intake during ICU stay
Changes in Resting Energy Expenditure (REE) measured with indirect calorimetry | All REE measurements during the ICU stay, recorded daily from ICU admission to ICU discharge, up to 52 weeks
  Changes in Resting Energy Expenditure (REE)

CONTACTS AND LOCATIONS:
Locations (1):
- Gelderse Vallei Hospital, Ede, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: V2 (2025-10-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT07312708/Prot_SAP_000.pdf